CLINICAL TRIAL: NCT04732091
Title: High Ultrasound Mechanical Index and MicrobuBBLEs to Reduce Acute Myocardial Infarction Burden I
Brief Title: Therapeutic Use of Contrast Ultrasound in Acute Coronary Artery Disease
Acronym: HUBBLE-I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Principal Investigator, Wilson Mathias Junior, Director Echocardiography Laboratory - Heart Institute, University of Sao Paulo General Hospital
Other Study IDs: 2018/06387-8
Record Dates: First submitted 2021-01-22; First posted 2021-02-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Acute Myocardial Infarction; Unstable Angina
Keywords: Ultrasound; Sonothrombolysis; Contrast agents; Microbubbles; Microvascular obstruction
MeSH Terms: conditions — Angina, Unstable | interventions — Ultrasonic Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Subproject 1 - acute STEMI: Participants with acute STEMI will receive intravenous infusion of microbubbles (3% Definity) with therapeutic ultrasound with 4-20 usec and custom designed high mechanical index (MI) impulses (1.1 to 1.3 MI) designed for the 1.8 MHz S5-1 transducer while waiting for percutaneous coronary intervention. Treatment will continue after procedure until complete a total of 50 minutes.
  Interventions: Procedure: Therapeutic ultrasound with 20 usec
- Subproject 2 - acute STEMI initially treated with fibrinolytic: Participants with acute STEMI initially treated with fibrinolytic therapy within 12 hours will receive intravenous infusion of microbubbles (3% Definity) with therapeutic ultrasound with 4-20 usec and custom designed high mechanical index (MI) impulses (1.1 to 1.3 MI) designed for the 1.8 MHz S5-1 transducer while waiting for percutaneous coronary intervention. A control group (PCI only) undergoing low MI (<0.2) imaging only with limited (no more than 3) diagnostic high MI impulses to assess regional wall motion and microvascular perfusion before and after PCI; High MI will continue after PCI procedure until complete a total of 50 minutes.
  Interventions: Procedure: Therapeutic ultrasound with 20 usec
- Subproject 3 - NSTEMI: Participants with NSTEMI or with high-risk unstable angina will receive intravenous infusion of microbubbles (3% Definity) with therapeutic ultrasound with 4-20 usec and custom designed high mechanical index (MI) impulses (1.1 to 1.3 MI) designed for the 1.8 MHz S5-1 transducer while waiting for percutaneous coronary intervention. A control group (PCI only) undergoing low MI (<0.2) imaging only with limited (no more than 3) diagnostic high MI impulses to assess regional wall motion and microvascular perfusion before and after PCI. High MI will continue after PCI procedure until complete a total of 50 minutes.
  Interventions: Procedure: Therapeutic ultrasound with 20 usec
- Subproject 4 - No reflow: Participants with acute STEMI will receive intravenous infusion of microbubbles (3% Definity) with therapeutic ultrasound with 4-20 usec and custom designed high mechanical index (MI) impulses (1.1 to 1.3 MI) designed for the 1.8 MHz S5-1 transducer while waiting for percutaneous coronary intervention. A control group (PCI only) undergoing low MI (<0.2 MI) imaging only with limited (no more than 3) diagnostic high MI impulses to assess regional wall motion and microvascular perfusion before and after PCI. High MI will continue after PCI procedure until complete a total of 50 minutes.
  Interventions: Procedure: Therapeutic ultrasound with 20 usec
- Subproject 6 - Pre-hospital care (ambulance): Participants with acute STEMI routing from the ambulance to the emergency department will receive intravenous infusion of microbubbles (3% Definity) with therapeutic ultrasound with 4-20 usec and custom designed high mechanical index (MI) impulses (1.1 to 1.3 MI) designed for the 1.8 MHz S5-1 transducer while waiting for percutaneous coronary intervention. A control group (PCI only) undergoing low MI (<0.2) imaging only with limited (no more than 3) diagnostic high MI impulses to assess regional wall motion and microvascular perfusion before and after PCI. High MI will continue after PCI procedure until complete a total of 50 minutes.
  Interventions: Procedure: Therapeutic ultrasound with 20 usec

INTERVENTIONS:
Procedure: Therapeutic ultrasound with 20 usec — A custom designed high mechanical index (MI) impulses at 4-20 usec and >1.0 mechanical index designed for the 1.8 MHz S5-1 transducer

SUMMARY:
Preclinical studies have demonstrated that high mechanical index (MI) impulses from a diagnostic ultrasound (DUS) transducer during an intravenous microbubble infusion (sonothrombolysis) can restore epicardial and microvascular flow in acute ST-segment elevation myocardial infarction (STEMI). The investigators propose to demonstrate the clinical effectiveness of sonothrombolysis in multiple centers and in a wide scenario of acute coronary syndromes.

DETAILED DESCRIPTION:
Initial safety and feasibility human studies demonstrated that intermittent high MI aimed at the myocardial microcirculation could improve capillary blood flow within the risk area and epicardial recanalization rates. In light of this, the investigators published the first prospective randomized human study showing the added value of sonothrombolysis to percutaneous coronary intervention (PCI). Sonothrombolysis improved recanalization rates and reduced infarct size, leading to sustained improvements in systolic function after STEMI. Since both diagnostic ultrasound and intravenous infusions of microbubbles are Class I indication to assess regional and global left ventricular function and risk area in patients with STEMI, the purpose of this study is to 1) demonstrate the clinical effectiveness of sonothrombolysis in multiple centers and in a wide scenario of acute coronary syndromes including pre-hospital care setting; and 2) develop a portable non-imaging ultrasound device prototype, simple-to-handle and capable of generating intermittent ultrasound pulses for sonothrombolysis.

A total of 540 subjects will be included in this study. Subjects will be randomized to either receive DUS guided high MI impulses within and outside the risk area during a continuous infusion of intravenous 3% Definity® or placebo. Comparisons between the two groups will be made on door to dilation times, survival, angiographic recanalization rates at initial angiography and reduction in microvascular obstruction and in infarct size determined by the salvageability index at cardiac magnetic resonance imaging (MRI) post-STEMI and using myocardial perfusion imaging. The effect of high-energy ultrasound therapy and microbubbles on the outcome of sympathetic hyperactivation and autonomic imbalance after MI will be also evaluated. Cardiac remodeling assessed by left atrial and ventricular volumes indexes and myocardial strain imaging will also be measured. Overall survival defined as the time from the start of treatment to death from any cause as well as new MIs events will be assessed.

The study will be divided into 6 subprojects: subproject 1 (n=70 in each group) - safety and efficacy of the therapeutic use of intermittent high-energy ultrasound and microbubbles in the recanalization of acute STEMI treated with primary PCI. Additionally, the investigators will assess the effect of sonothrombolysis on autonomic function, cardiac function and intracellular signaling. All patients will receive conventional PCI approach, including aspirin 325 milligram, clopidogrel 600 milligrams and heparin bolus (5000 units), followed by primary PCI using glycoprotein 2b/3a inhibitors as anti-thrombotic agents using established protocols. Besides angiographic recanalization rates at the time of presentation to the catheterization laboratory, participants will have a fully echocardiography study including myocardial perfusion imaging and strain imaging, serum microRNAS for detecting endothelial cells shear-stress and autonomic control assessment (heart rate and systolic blood pressure variability) at the baseline, 72-96 hours, 30 days and 6 months of follow up. A iodine-123 meta-iodobenzylguanidine (MIBG) cardiac scintigraphy will be carried out at 30 days and 6 months follow up, and exercise echocardiogram at 6 months. Subproject 2 (n=70 in each group) - safety and efficacy of the therapeutic use of intermittent high-energy ultrasound and microbubbles in the recanalization of acute STEMI in patients initially treated in a primary hospital with fibrinolytic therapy within 12 hours. Angiographic recanalization rates at initial angiography and in infarct size determined by the salvageability index at cardiac MRI post-STEMI, and cardiac death and a new MI episode are the main objectives. Participants will receive STEMI/PCI treatment as per current guidelines using standard protocols similar to subproject 1. In addition, both groups will undergo elective PCI after fibrinolytic therapy. Besides angiographic recanalization rates at the time of presentation to the catheterization laboratory, a comprehensive echocardiography study including myocardial perfusion and strain imaging, MRI and exercise echocardiogram will be performed at the time of presentation and during 72-96 hours, 30 days, 3 months and 6 months of follow up. Subproject 3 (n=70 in each group) - safety and efficacy of the therapeutic use of intermittent high-energy ultrasound and microbubbles in the recanalization of acute myocardial infarction without segment elevation or with high-risk unstable angina (NSTEMI). Subjects presenting without persistent ST-segment elevation acute coronary syndromes undergoing early invasive strategy within 24 hours will be randomized to either receive diagnostic ultrasound guided high MI impulses during a continuous infusion of intravenous 3% Definity® or placebo. Participants will receive conventional medical treatment, including aspirin 325 milligram, clopidogrel 600 milligrams and unfractionated heparin weight-adjusted iv. bolus or in combination with glycoprotein 2b/3a inhibitors followed by primary PCI using established protocols as per current guidelines. A comprehensive echocardiography study including myocardial perfusion echocardiography and exercise echocardiogram will be carried out at the baseline, 72-96 hours, 30 days- and 6 months of follow up. Subproject 4 (n=30 in each group): safety and efficacy of the therapeutic use of intermittent high-energy ultrasound and microbubbles in reducing microvascular obstruction and myocardial infarction size after primary PCI in patients with anterior wall myocardial infarction. Participants will receive STEMI/PCI approach as per guidelines likewise subprojects 1 and 2. In order to assess microvascular obstruction and no reflow phenomenon, a comprehensive echocardiography study, including myocardial perfusion imaging and myocardial strain will be performed at baseline, 2 months and 6 months of follow up. MRI will be performed at 3 days and 3 months of follow up. Subproject 5: this subproject will be dedicated to the development of an automated hands-free portable prototype emitting ultrasound waves of intermittent high-energy capable of promoting sonothrombolysis. Subproject 6 (n=30 in each group): a pilot study on the therapeutic use of intermittent high-energy ultrasound and microbubbles in the recanalization of acute STEMI in the pre-hospital setting (ambulances). Subjects with acute STEMI will be randomized to either receive diagnostic ultrasound guided high MI impulses during a continuous infusion of intravenous 3% Definity® or placebo while routing from the ambulance to the emergency department. At the admission hospital, all patients will receive conventional PCI approach, including aspirin 325 milligram, clopidogrel 600 milligrams and heparin bolus (5000 units), followed by primary PCI using glycoprotein 2b/3a inhibitors as anti-thrombotic agents using established protocols as per aforementioned subprojects. A complete echocardiography study including myocardial perfusion and strain, and exercise echocardiogram will be carried out at baseline, 72-96 hours, 30 days- and 6 months of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥30 years with STEMI with less than 12 hours of chest pain onset.
* Age ≥30 years with STEMI initially treated in a primary setting by fibrinolytic therapy within 12h
* Age ≥30 years with NSTEMI with high-risk unstable angina who will undergo elective PCI
* Eligible for emergent PCI therapy.
* No contraindications or hypersensitivities to ultrasound contrast agents

Exclusion Criteria:

* Known or suspected hypersensitivity to ultrasound contrast agent used for the study.
* Cardiogenic Shock.
* Life expectancy of less than two months or terminally ill.
* Known bleeding diathesis or contraindication to glycoprotein 2b/3a inhibitors, anticoagulants, or aspirin.
* Known large right to left intracardiac shunts or severe pulmonary hypertension.
* Patients who received thrombolytic therapy previously to enrollment.
* Women of childbearing potential.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ST elevation myocardial infarction (STEMI) with less than 12 hours of chest pain onset, STEMI initially treated with fibrinonilytic therapy, NSTEMI or high-risk angina undergoing early invasive PCI, anterior wall (LAD territory) acute STEMI, and acute STEMI with less than 12 hours of chest pain onset in the pre-care setting (ambulance) eligible for emergent percutaneous coronary intervention therapy.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Angiographic recanalization rate | At initial angiography
  Percentage of patients with acute STEMI and open artery at initial angiography (TIMI I)

SECONDARY OUTCOMES:
Salvageability index | 72-96 hours and 3 months post infarction
  Percentage of myocardium with viability within the risk area obtained by magnetic resonance imaging
Overall survival | 30 days post infarction
  The time from the start of treatment to death from any cause
Cardiac remodeling | 72-96 hours, 30 days and at 6 months
  Left ventricular and left atrial volumes (mL) will be measured using comprehensive two-dimensional echocardiography
Myocardial Mechanics | 72-96 hours, 30 days and at 6 months
  Percentage of myocardial deformation (%), ie. left ventricular strain imaging will be assessed to detect subclinical myocardial dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Mathias Jr, MD, PhD, Principal Investigator — Heart Institute - University of São Paulo Medical School; Jeane Tsutsui, MD, PhD, Principal Investigator — Heart Institute - University of São Paulo Medical School; Thomas R Porter, MD, Principal Investigator — University of Nebraska Medical Center, Omaha, NE
Locations (2):
- Department of Internal Medicine, Division of Cardiovascular Medicine, University of Nebraska Medical Center, Omaha, Nebraska, United States
- Heart Institute of Clinical Hospital of Medical School of University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The data will be saved into a research encrypted platform available only to study group researchers. Participants will be non-identifiable and results will be blinded to reviewers. The platforms included are RedCap and Castor.